CLINICAL TRIAL: NCT07403422
Title: Effects of Forward Head Posture on Cervical Proprioception, Muscle Endurance, and Cardiopulmonary Function During Cognitive-Motor Tasks Among University Students: A Cross-Sectional Study
Brief Title: Effects of Forward Head Posture on Cervical Proprioception, Muscle Endurance, and Cardiopulmonary Function During Cognitive-Motor Tasks Among University Students
Status: Completed | Type: Observational
Sponsor: Abeer Abdrabo (Other)
Responsible Party: Sponsor-Investigator, Abeer Abdrabo, Lecture, Department of Neuromuscular Disorder, Faculty for Physical Therapy, Cairo University, Cairo, Egypt, Isra University, Jordan
Organization: Isra University, Jordan (Other)
Other Study IDs: [NO.P.T/REC/230010/4/12/2023]]
Record Dates: First submitted 2026-01-18; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Forward Head Posture

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group / Cohort 1 Group Name: Forward Head Posture Group: This cohort includes participants diagnosed with forward head posture based on standardized postural assessment criteria.
  Interventions: Other: No intervention
- Group / Cohort 2 Group Name: Normal Head Posture (Control) Group: This cohort includes participants with normal head and neck posture and no musculoskeletal or neurological disorders.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Forward head posture is commonly observed among university students and may influence cervical sensorimotor function and physiological responses during functional activities. The purpose of this observational cross-sectional study is to examine the association between forward head posture and cervical proprioception, deep cervical muscle endurance, and cardiopulmonary responses during a cognitive-motor task in university students.

DETAILED DESCRIPTION:
This is an observational cross-sectional study conducted among healthy university students aged 18 to 26 years. The study aims to investigate the relationship between forward head posture and cervical joint position sense, deep cervical muscle endurance, and cardiopulmonary responses during a combined cognitive-motor task. No therapeutic intervention or treatment is applied.

ELIGIBILITY:
Inclusion Criteria:

* University students aged 18 to 26 years
* Both male and female participants
* Apparently healthy individuals
* Ability to understand and follow study instructions
* Willingness to participate and provide written informed consent

Exclusion Criteria:

* Age below 18 years or above 26 years
* History of cervical spine surgery or cervical fracture
* Presence of neurological disorders affecting the cervical spine or balance
* Chronic cardiopulmonary diseases
* Current or recent neck or shoulder pain within the past 6 months
* Any musculoskeletal condition that may affect cervical posture or movement

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of healthy male and female university students aged 18 to 26 years, recruited from the university campus. Participants represent a young adult population without known neurological, musculoskeletal, or cardiopulmonary conditions that could influence cervical posture or sensorimotor performance.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2025-11-14 (Actual); Primary Completion 2026-01-07 (Actual); Study Completion 2026-01-10 (Actual)

PRIMARY OUTCOMES:
Cervical joint position error measured using a smartphone-based inclinometer | At baseline
  Cervical proprioception will be assessed by measuring joint position error (JPE) during cervical flexion, extension, and rotation using a smartphone-based inclinometer. Participants will attempt to reposition their head to a neutral target position with eyes closed. The absolute repositioning error (in degrees) will be calculated, and the mean JPE will be used for analysis.

SECONDARY OUTCOMES:
Deep cervical flexor endurance measured by the craniocervical flexion endurance test | At baseline
  Deep cervical flexor endurance will be assessed using the craniocervical flexion endurance test. Participants will perform a chin-tuck head lift in the supine position and hold the position as long as possible. Endurance time will be recorded in seconds.
Cervical extensor endurance measured by a cervical extensor endurance test | At baseline
  Cervical extensor muscle endurance will be assessed using a cervical extensor endurance test in the prone position. Participants will maintain the head in a neutral horizontal position for as long as possible. Endurance time will be recorded in seconds.
Heart rate measured during a cognitive-motor dual-task using a chest-strap heart rate monitor | During a single 3-minute cognitive-motor task session
  Heart rate will be recorded during a combined stepping and cognitive subtraction task using a validated chest-strap heart rate monitor. The mean heart rate during the task will be used for analysis.
Respiratory rate measured during a cognitive-motor dual-task | During a single 3-minute cognitive-motor task session
  Respiratory rate will be measured during the same cognitive-motor dual-task by counting breaths per minute. The mean respiratory rate during the task will be used for analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, Aqaba, Jordan

IPD SHARING:
Plan to Share IPD: No
"Individual participant data (IPD) will not be shared to protect the privacy and confidentiality of university students. The data include sensitive health and physical measurements, and sharing them could risk identification of participants despite de-identification efforts. Additionally, no formal data-sharing agreements are in place."